CLINICAL TRIAL: NCT05602948
Title: ACTIVE SCHOOL - Effects on Academic Performance of Novel Approaches to Increase Physical Activity in School-children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College Copenhagen (Other)
Collaborators: University of Copenhagen (Other); UCL University College, Denmark (Other)
Responsible Party: Principal Investigator, Anna Bugge, Associate Professor (Docent), University College Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Alias: 200511110
Record Dates: First submitted 2022-10-25; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Academic Performance
Keywords: Physical activity; Embodied cognition; Mathematics; Reading
MeSH Terms: conditions — Motor Activity | interventions — Jogging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 'Run, Jump & Fun' intervention (Experimental): The "Run, jump & fun" intervention consists of four 30 minutes sessions per week for one school year. Activities are mostly conducted as whole class activities. Head of schools and teachers/school pedagogues are involved in an initial intervention establishing process, guided by Active School personnel. The aim is to create a local plan for the intervention tailored to the particular school. Examples are "movement band", structured activities during recess with older students (13-15 years olds), etc. Activities are created to be fun, motivating and with moderate to high intensity PA.
  Interventions: Behavioral: 'Run, Jump & Fun' intervention
- 'Move & Learn' intervention (Experimental): This intervention is implemented as PA for 30 min in two Mathematics and two Danish lessons each week for one school year. Activities are conducted at whole-class level.
  The physical activities in "Move & Learn" are closely linked to the Mathematic curriculum and the Danish curriculum. The way the body is integrated in the learning task can vary. Examples are bodily or motor-skill demanding activities or less vigorous activities, e.g. standing up miming, using hand gestures or facial expressions. An important aspect of the interventions is that movements should be task relevant. The intervention is developed based on the embodied learning theory.
  Interventions: Behavioral: 'Move & Learn' intervention
- Control (No Intervention): Control schools will continue their usual practice.

INTERVENTIONS:
Behavioral: 'Run, Jump & Fun' intervention — The intervention can be designed e.g. to consist of morning sessions each schoolday (except days with PE) or with different time slots at different weekdays. Activities are mainly conducted by school personnel, but can be supplemented by activity sessions during recess once a week lead by older students. Further, to create variation and inspire teachers, external PA parties, for example instructors from local sports clubs are invited to conduct sessions for the students and deliver teaching materials.
  To align with the aim of the Danish school system, activities must have a pedagogical purpose.
  Both the "Run, jump & fun" and the "Move & learn" interventions have a set of strategies underpinning implementation (see Move & Learn" for more details).
  Both interventions will be grounded in Self-Determination Theory and all activities will be designed to be motivating and enjoyable for all children including those neither particularly fit nor enthusiastic about PA.
  Arms: 'Run, Jump & Fun' intervention
Behavioral: 'Move & Learn' intervention — The physical activities in "Move & Learn" are closely linked to the subject curricula. The bodily integrating in the learning task can vary between high bodily engagement and less demanding activities.
  Both the "Run, jump & fun" and the "Move & learn" interventions have a set of strategies underpinning implementation. These strategies include; 1) Initial workshops and follow-up courses for school personnel to ensure ownership, empowerment and knowledge in order to implement the interventions, 2) Teaching materials and resources, like posters, booklets etc., 3) A set of core principles for the two different interventions to ensure that the interventions are implemented as intended, and 4) Mandatory school meetings for staff and heads to ensure motivation.
  Both interventions will be grounded in Self-Determination Theory and all activities will be designed to be motivating and enjoyable for all children including those neither particularly fit nor enthusiastic about PA.
  Arms: 'Move & Learn' intervention

SUMMARY:
The overall aim of ACTIVE SCHOOL is to investigate the effects of two different physical activity (PA) interventions on academic performance (AP), cognition, wellbeing, health and motivation. The two different approaches to PA in schools are based on;

1. 'Embodied cognition' focusing on fine and gross motor PA closely related and highly relevant to the learning task. 'Embodied cognition' builds upon theory suggesting that movement and performing actions leads to the construction of enhanced mental representations e.g. strengthening memory recall. This intervention is called 'MOVE & LEARN'.
2. 'Exercise and cognition theory focusing mainly on gross motor movements (e.g. aerobic exercise) which is not relevant to the learning task and with no temporal connection to the learning task. The assumed positive effects are explained by physiological adaptations leading to changes in cognition, which potentially can affect AP. This intervention is called 'RUN, JUMP & FUN'.

Based on this, the aims of ACTIVE SCHOOL are to develop two types of school-based PA interventions in close collaboration with the participating teachers, students and schools AND to investigate the effects of these two interventions on AP in a large school-based cluster-RCT with an intervention length of one school year.

The ACTIVE SCHOOL study consists of three phases: Phase 1) Development of the intervention, Phase 2) Pilot testing and, Pase 3) A three-armed randomized controlled trial (RCT). Participants will be students in 3rd grade (8-10 years-old) and their teachers/school pedagogues.

The development phase started in August 2021 and is still ongoing. The pilot study will run in September-November 2022 and the RCT from August 2023 to June 2024. In the RCT, schools will be randomly allocated to one of three intervention/control arms: 1) 'MOVE & LEARN', 2) 'RUN, JUMP & FUN' or 3) control. Primary and secondary outcomes will be collected before and after the intervention period to assess the intervention effects. Both the pilot and RCT study has been granted approval by the local ethics committee, and all rules from the Danish Data Protection Agency and GDPR will be followed. The RCT study will follow the Consolidated Standards of Reporting Trials (CONSORT) guidelines for RCT studies.

ELIGIBILITY:
Inclusion Criteria:

* Children in 3rd grade

Exclusion Criteria:

* Children with cognitive or physical disabilities hindering participation in the project activities

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1200 (Estimated)
Dates: Start 2021-01-02 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Mathematics performance by standardized national tests. Average of three domains (algebra, geometry, and basic mathematics skills) | Change from baseline Mathematics performance at 10 months
  Danish National Test System. The tests are computerized and composed in a progressive manner, depending on the individual child's performance, such that correct answers lead to more difficult subsequent questions, and incorrect answers lead to easier subsequent questions. The final test result is therefore based on the level of difficulty, not the number of correct answers. The tests are divided into three different domains; for mathematics: algebra, geometry, and basic mathematics skills. No aids are permitted during the tests. The tests are scored on a scale from 0 to 100 in each domain. For this study, the mean of the three domains will be used for analyses

SECONDARY OUTCOMES:
Reading performance by standardized tests | Change from baseline reading performance at 10 months
  Hogrefe Psykologisk Forlag. (2014).
Executive functions measured by a digit span test and a spatial working memory test (SWM) which assess working memory and attention | Change from baseline executive function measures at 10 months
  WAIS-IV Administration and Scoring Manual. San antonio, TX: Psychological Corporation (2008) and Spatial Working Memory (SWM) | Cambridge Cognition. https://www.cambridgecognition.com/cantab/cognitive-tests/executive-function/spatial-executive-function-swm/.
Objective PA measurements by accelerometry for one week | Change from baseline objective PA measurements at 10 months
  ActiGraph GT3X+, LLC, Pensacola, Florida, USA
Cardiorespiratory fitness using a validated modified shuttle run test | Change from baseline cardiorespiratory fitness at 10 months
  Andersen, L. B., Andersen, T. E., Andersen, E. & Anderssen, S. A. An intermittent running test to estimate maximal oxygen uptake: the Andersen test. J. Sport. Med. Phys. Fit. 48, 434-437 (2008)
Anthropometry (stature, body mass, waist circumference and puberty status) | Change from baseline anthopometry measures at 10 months
  Tanner, J. M. Growth and maturation during adolescence. Nutr. Rev 39, 43-55 (1981).
Register data on socioeconomic status (SES) and education of parents | Baseline
  Danmarks_Statistik. Data for research, Statistics Denmark. Research data (2019
Questionnaires (parental health, diseases diagnosed in the participating children, sleep, diet) | Baseline
  Custom made
Questionnaire of quality of life | Change from baseline Kidscreen-27 at 10 months
  The KIDSCREEN-27 quality of life measure for children and adolescents: psychometric results from a cross-cultural survey in 13 European countries. Quality of life research. vol. 16 1347-1356 (2007).
Questionnaire of intrinsic motivation and feeling of enjoyment, competence, autonomy and relatedness | Change from baseline Intrinsic Motivation Inventory at 10 months
  Self-Determination. Intrinsic Motivation Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Bugge, PhD, Principal Investigator — University College Copenhagen
Locations (1):
- University College Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Jeppesen LS, Damsgaard L, Stolpe MN, Melcher JNS, Wienecke J, Nielsen G, Smedegaard S, Henriksen AH, Hansen RA, Hillman CH, Tammelin TH, Resaland GK, Daly-Smith A, Bugge A. Study protocol for the ACTIVE SCHOOL study investigating two different strategies of physical activity to improve academic performance in Schoolchildren. BMC Pediatr. 2024 Mar 9;24(1):174. doi: 10.1186/s12887-024-04647-9. PMID 38461348